CLINICAL TRIAL: NCT01004445
Title: A Double-Blind, Placebo-controlled Parallel Group, Phase II Dose-Ranging Study of Nebulized Amikacin Delivered Via the Pulmonary Drug Delivery System (PDDS) in Ventilated Patients With Nosocomial Pneumonia Due to Gram Negative Organisms
Brief Title: A Study to Determine the Correct Dose of Amikacin Which is Delivered Directly to the Lungs of Ventilated Patients as an Aerosol Via an Investigational Device Called the Pulmonary Delivery Device System (PDDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMIK-04-02
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Pneumonia
Keywords: Pneumonia; Adjunctive treatment; Gram-negative bacteria
MeSH Terms: conditions — Pneumonia | interventions — Amikacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Amikacin (BAY41-6551)
- Arm 2 (Experimental)
  Interventions: Drug: Amikacin (BAY41-6551)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amikacin (BAY41-6551) — Single daily dose of 400 mg aerosolized amikacin and a single dose of aerosolized placebo on a rotating every 12hr schedule
  Arms: Arm 1
Drug: Amikacin (BAY41-6551) — Daily dose of 800 mg aerosolized amikacin delivered in two divided doses of 400 mg per aerosol treatment every 12hr
  Arms: Arm 2
Drug: Placebo — Two aerosol treatments per day (one treatment every 12hr)
  Arms: Arm 3

SUMMARY:
This study is part of a research program too see if amikacin delivered as an aerosol directly to the lungs in combination with IV antibiotic therapy can help intubated patients with gram-negative pneumonia get better faster than when given intravenous antibiotics alone. The primary purpose of this study is to determine the correct dose of amikacin which is delivered directly to the lungs as an aerosol via an investigational device called the Pulmonary Delivery Device System (PDDS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older with a clinical diagnosis of VAP, HAP or HCAP who are expected to be on mechanical ventilation for at least 3 days

Exclusion Criteria:

* Patients with compromised of suppressed immune systems, severe hypoxemia, PEEP>15cm H2O, creatinine>2 mg/dL, or who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-05; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve a C(max) for amikacin in tracheal aspirates at least 25 times greater than the reference MIC for hospital-acquired organisms and an AUC (0-24 hr) / MIC ratio that is 100 or greater on Day 1 | Day 1

SECONDARY OUTCOMES:
Mean C(max) and mean AUC of amikacin in tracheal aspirates | Day 1 and Day 3 of treatment period
Mean ratio of C (max) / MIC and mean ratio of AUC (0-24 hr) / MIC | Day 1 and Day 3 of treatment period
Clinical cure rate | Test of cure visit (7 days post last treatment dose)
Microbiological eradication rate of identified pathogens | Test of cure visit (7 days post last treatment dose)
Microbiological persistence rate | Test of cure visit (7 days post last treatment dose)
New infection rate | Test of cure visit (7 days post last treatment dose)
Assessment of adverse events related to drug or device | Treatment period, early post treatment period, test of cure visit, and late post treatment
Assessment of abnormal laboratory values | Treatment period, early post treatment period, test of cure visit, and late post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- United States (7):
  - Birmingham, Alabama
  - Melbourne, Florida
  - Albany, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Houston, Texas
  - San Antonio, Texas
- France (4):
  - Angers
  - Limoges
  - Paris
  - Rouen
- Spain (3):
  - Barcelona
  - Madrid
  - Murcia

REFERENCES:
- [Derived] Niederman MS, Chastre J, Corkery K, Fink JB, Luyt CE, Garcia MS. BAY41-6551 achieves bactericidal tracheal aspirate amikacin concentrations in mechanically ventilated patients with Gram-negative pneumonia. Intensive Care Med. 2012 Feb;38(2):263-71. doi: 10.1007/s00134-011-2420-0. Epub 2011 Dec 7. PMID 22147112